CLINICAL TRIAL: NCT02786758
Title: Eliminating Hepatitis C Transmission by Enhancing Care and Treatment Among HIV Co-infected Individuals: The Co-EC Study
Brief Title: Eliminating Hepatitis C Transmission by Enhancing Care and Treatment Among HIV Co-infected Individuals
Acronym: co-EC
Status: Completed | Type: Observational
Sponsor: Macfarlane Burnet Institute for Medical Research and Public Health Ltd (Other)
Collaborators: The Alfred (Other)
Responsible Party: Sponsor
Other Study IDs: burnet_coec_2016
Record Dates: First submitted 2016-05-03; First posted 2016-06-01 (Estimated); Last update posted 2020-02-28 (Actual); Status verified 2020-02

CONDITIONS: Hepatitis C; HIV
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Standard of care blood tests (whole blood) will be obtained at screening and subsequent visits, depending on HCV medication regimen and health status, in order to assess: HCV genotype, HCV RNA viral load, host IL28B genotype, liver function, full blood examinations, iron studies, vitamin D, lipid profile, clotting profile, alpha-feto protein, HIV RNA viral load and hepatitis B virus serology. In addition, a study specimen for HCV NS3/NS5 sequencing will be collected at screening and stored. Specimens for pregnancy tests will be collected where applicable. Biospecimens from this study will be frozen and stored in secure laboratories at the Burnet and Victorian Infectious Diseases Reference Laboratory, for a minimum of 15 years in a biobank, under custody of the principal investigator.
Oversight: Data Monitoring Committee: Yes

SUMMARY:
This study will offer proof of concept that scaling up treatment for Hepatitis C virus (HCV) in individuals co-infected with HIV could lead to elimination of HCV/HIV co-infection in gay and bisexual men by treating prevalent infection, thereby reducing new primary infections and re-infection.

DETAILED DESCRIPTION:
The co-EC study aims to to enhance HCV care and treatment among HIV-infected individuals through a predominantly nurse-led model of care in primary care as well as hospital settings. It involves:

1. A nurse-led model of care in primary health care to increase access to PBS HCV treatment with interferon-free HCV antiviral treatment; and
2. An integrated HCV/HIV surveillance system and database to deliver and monitor the impact of the program at the local and statewide level.

The study is based in Victoria, Australia where the highest prevalence of HIV/HCV co-infection is in gay and bisexual men (GBM). HCV infection is a significant health issue among individuals with HIV infection and has been associated with more rapid progression to HCV-related liver disease and increased risk for cirrhosis and liver cancer. Hepatitis C is a major cause of hospital admissions and is a leading cause of death among HIV-infected persons.

The advent of directly acting antiviral (DAA) treatment provides us with a unique opportunity to increase the number of people accessing hepatitis C treatment. Importantly it is likely that the treatment could be administered in the primary health care setting improving treatment capacity and accessibility, whilst potentially reducing treatment costs.

The primary objectives of co-EC Study are:

1. Achieve HCV sustained virological response (SVR12) to treatment among HIV co-infected participants in a real-world primary care or hospital clinic setting; and
2. Measure the impact of treating HCV in HIV infected individuals on primary HCV and reinfection incidence and HCV prevalence in gay and bisexual men in Victoria.

The study design involves an open label, non-randomised clinical trial of hepatitis C treatment for people with HIV coinfection. Treatment will involve any combination of hepatitis C antiviral therapy approved for use in Australia appropriate for the participants' hepatitis C genotype and selected at the decision of their treating clinicians.

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 years;
2. Attendance for medical care of HIV at any study site;
3. Evidence of chronic HCV infection (HCV antibody or RNA positive for ≥6 months and HCV RNA positive);
4. HIV infected;
5. Willing and able to provide written informed consent;

Subjects must meet routine clinical care criteria for commencing HCV treatment, in accordance with Australian licensing, prescribing restrictions, manufacturers' recommendations and best- practice clinical care.

Exclusion Criteria:

1. Pregnancy or breastfeeding at time of HCV antiviral treatment;
2. Evidence of any condition, therapy, laboratory abnormality or other circumstance (current or prior) that may confound the study's results, or interfere with participation for the full duration of the study, such that it is not in the best interest of the participant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Any HCV/HIV co-infected individuals attending any of the six clinical sites involved in this study will be eligible to participate. While the study's objective are to focus on HCV among HIV infected gay and bisexual men, females and men not identifying as gay or bisexual will also be able to participate and receive HCV treatment.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2019-07 (Actual); Study Completion 2019-08 (Actual)

PRIMARY OUTCOMES:
Treatment uptake | 18 months
  The number of individuals receiving at least one dose of HCV treatment among all HCV/HIV coinfection individuals in care (seen within the previous 12 months) at that health service.
Sustained virological response after treatment (SVR12) | Change in sustained viral response rates post-treatment (SVR12).
  Determined using any licensed qualitative HCV RNA test among all those receiving at least one dose of HCV treatment.
HCV prevalence | 12 months
  The proportion HCV RNA positive of all HIV infected individuals in care (seen within the previous 12 months) at that health service. Statewide HCV prevalence will be determined as a proportion of all HIV infected individuals in care (determined by at least one HIV RNA within the previous 12 months).
HCV incidence | 12 months
  The number of newly detected HCV RNA cases occurring among all HIV infected individuals during the time in care (determined by clinical visit or HIV RNA test within the previous 12 months).

SECONDARY OUTCOMES:
Change in HCV testing among HIV-infected gay and bisexual men | 18 months
  Hypothesized that primary care and clinic-based nurses will increase the proportion of people in care receiving HCV testing annually and repeat testing at intervals recommended by national guidelines.
Change in number of HIV/HCV infected gay and bisexual men who have a complete management plan including HCV RNA status, FibroScan and liver function tests. | 18 months
  Number of HCV/HIV reinfections in gay and bisexual men management plan will be increased.
Medical adherence | Up to 24 weeks, documented at each study visit
  Primar care and clinic based nurses will increase medical adherence.

CONTACTS AND LOCATIONS:
Overall Officials: Margaret Hellard, Principal Investigator — Burnet Institute; Joseph Doyle, Principal Investigator — The Alfred
Locations (6):
- Australia (6):
  - Melbourne Sexual Health Centre, Carlton, Victoria
  - Northside Clinic, Fitzroy North, Victoria
  - Alfred Health, The Alfred Hospital, Melbourne, Victoria
  - Melbourne Health, Royal Melbourne Hospital, Parkville, Victoria
  - Prahran Market Clinic, Prahran, Victoria
  - Centre Clinic, St Kilda, Victoria

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Doyle JS, van Santen DK, Iser D, Sasadeusz J, O'Reilly M, Harney B, Traeger MW, Roney J, Cutts JC, Bowring AL, Winter R, Medland N, Fairley CK, Moore R, Tee BK, Asselin J, El-Hayek C, Hoy JF, Matthews GV, Prins M, Stoove MA, Hellard ME. Microelimination of Hepatitis C Among People With Human Immunodeficiency Virus Coinfection: Declining Incidence and Prevalence Accompanying a Multicenter Treatment Scale-up Trial. Clin Infect Dis. 2021 Oct 5;73(7):e2164-e2172. doi: 10.1093/cid/ciaa1500. PMID 33010149